CLINICAL TRIAL: NCT00955591
Title: Comparison of Flocked vs. Dacron Swab for Anal Cytology, Correspondence With High Resolution Anoscopy
Brief Title: Comparing Two Types of Swabs in Collecting Cell Samples for Anal Pap Tests and Human Papillomavirus Tests in Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDR0000643881; UCLA-0901062; IRB# 09-01-062-02
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2016-09

CONDITIONS: Anal Cancer; Nonneoplastic Condition; Precancerous Condition
Keywords: human papilloma virus infection; anal cancer; HIV infection
MeSH Terms: conditions — Anus Neoplasms; Precancerous Conditions; Papillomavirus Infections; HIV Infections | interventions — Papanicolaou Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- swab test (Other)
  Interventions: Other: Papanicolaou test

INTERVENTIONS:
Other: Papanicolaou test

SUMMARY:
RATIONALE: Doctors use a swab to collect cell samples when testing for anal cancer and human papillomavirus. It is not yet known which type of swab is more effective in collecting cell samples for anal Pap tests and human papillomavirus tests in men who have sex with men.

PURPOSE: This clinical trial is comparing two types of swabs in collecting cell samples for anal Pap tests and human papillomavirus tests in men who have sex with men.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether the anal cytology screening outcome derived from specimens collected by a flocked nylon swab are equivalent to those derived from Dacron swab specimens in men who have sex with men.
* To determine whether the number and type-specific identification for human papillomavirus derived from specimens collected by a flocked nylon swab are equivalent to those derived from Dacron swab specimens.

OUTLINE: Dry sterile Dacron swabs and flocked nylon swabs are used to collect intra-anal cytology specimens for anal Pap testing and human papillomavirus typing. Participants undergo a digital rectal examination and high-resolution anoscopy. If lesions are identified, an anal biopsy is performed for histological examination.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected or -uninfected adult men who have sex with men
* Concurrent enrollment in the Multicenter AIDS Cohort Study required

Exclusion Criteria:

* history of anal perforation or other medical contraindications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-03-12 (Actual); Primary Completion 2011-12-12 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Comparison of anal cytology screening outcome derived from specimens collected by a flocked nylon swab vs a Dacron swab | a day

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Wiley, Ph.D. RN, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Wiley DJ, Hsu H, Bolan R, Voskanian A, Elashoff D, Young S, Dayrit R, Barman P, DeAzambuja K, Masongsong EV, Martinez-Maza O, Detels R. Comparison of 2 anal cytology protocols to predict high-grade anal intraepithelial neoplasia. J Low Genit Tract Dis. 2013 Oct;17(4):414-24. doi: 10.1097/LGT.0b013e318281d36e. PMID 23595039